CLINICAL TRIAL: NCT00362349
Title: A Single-arm, Open Label, Multi-centre Study Evaluating the Efficacy and Safety of Ig NexGen 10% in Patients With Idiopathic Thrombocytopenic Purpura (ITP)
Brief Title: Ig NextGen 10% in Idiopathic Thrombocytopenic Purpura (ITP) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSLCT-ITP-05-21
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2009-02

CONDITIONS: Idiopathic Thrombocytopenic Purpura (ITP)
Keywords: ITP; IVIg; Platelet count; Bleeding
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): IVIg
  Interventions: Drug: IgNextGen 10%

INTERVENTIONS:
Drug: IgNextGen 10% — Ig NextGen 10% is a liquid formulation and is to be administered intravenously. At the discretion of the Investigator, patients could be administered Ig NextGen 10% in accordance with either of two dosage regimens:
  Regimen One: 1 g/kg body weight of Ig NextGen 10% administered daily for two days.
  Regimen Two: 0.4 g/kg body weight of Ig NextGen 10% administered daily for five days

SUMMARY:
Idiopathic Thrombocytopenic Purpura (ITP) is an autoimmune bleeding disorder characterised by isolated low platelet counts. The aim of treating patients with ITP is to increase the platelet concentration and reduce the risk of bleeding. A number of controlled multi-centre studies have demonstrated that Intravenous Immunoglobulin (IVIg) therapy produces a rapid rise in platelet counts within a 24 to 72 hour period. This study will evaluate the efficacy and safety of Ig NextGen 10% in adult patients with ITP.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of ITP
* platelet count of <50 X 10^9

Exclusion Criteria:

* planned splenectomy
* previous non-responders to IVIg treatment
* known or suspected hypersensitivity or previous evidence of severe side effects to immunoglobulin therapy
* patients who have received treatment with:

  1. IVIg or anti-D immunoglobulin
  2. immunosuppressive, any other immunomodulatory drug(s) or other active treatment(s)for ITP within three weeks prior to first day of study drug administration
  3. patients who have received IV administration of steroids OR have had a change of oral corticosteroid treatment OR danazol within 15 days prior to first day of study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Efficacy | 90 days

SECONDARY OUTCOMES:
Safety | 97 days

CONTACTS AND LOCATIONS:
Overall Officials: Beng N/A Chong, Professor, Principal Investigator — The St George Hospital (NSW, Australia)
Locations (8):
- Australia (8):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - St George Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Redcliffe Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia